CLINICAL TRIAL: NCT03393533
Title: Evaluation of the Effectiveness of the Use of the Therapeutic Bandage Method in Third Molar Surgery. Splint-mouth Randomized Blind Controlled Clinical Trial
Brief Title: Evaluation of the Effectiveness of the Use of the Therapeutic Bandage Method in Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Michelle Bianchi de Moraes, Assistant Professor, Department of Diagnosis and Surgery, São Paulo State University (Unesp), Institute of Science and Technology, São José dos Campos, Brazil., Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Unesp
Record Dates: First submitted 2017-12-05; First posted 2018-01-08 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Pain
Keywords: Third molar;; Oral surgery;; Pain;; Edema;; Trismus.
MeSH Terms: conditions — Pain; Edema; Trismus

STUDY DESIGN:
Intervention Model Description: The sample will consist of 32 lower third molars, semi-inclusively or included. This study will be a randomized, blind, controlled, split-mouth clinical trial, divided into two groups simultaneously, namely:
  Group I (16 teeth) - without therapeutic banding on the face, after the third molar extraction.
  Group II (16 teeth) - with therapeutic banding on the face, after the third molar extraction.
Who Masked: Care Provider
Masking Description: Surgical procedures were always performed by the same surgeon and assistant, who was unaware of the group that belonged to the patient, as well as the patient himself. This randomization was performed involving numbers and envelopes, being only the investigator's knowledge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Other): Extraction third molar with pre and postoperative evaluation of edema, pain and trismus
  Interventions: Procedure: Group II
- Group II (Active Comparator): Extraction third molar with therapeutic bandage pre and postoperative evaluation of edema, pain and trismus
  Interventions: Procedure: Group I

INTERVENTIONS:
Procedure: Group I — Extraction third molar without the application of therapeutic bandaging in the face and with evaluation of edema, pain and trismus
  Arms: Group II
Procedure: Group II — Extraction third molar with the application of therapeutic bandaging in the face and with evaluation of edema, pain and trismus
  Arms: Group I

SUMMARY:
Extraction of lower third molars semi-included or included is one of the most performed procedures in oral surgery, and inherent to the procedure there is a postoperative inflammatory response. Among the factors most routine to this response are pain, edema and trismus. The therapy taping has advantages in its use in the physiotherapy of several specialities, leading to the correction of muscular functions, reduction of edema, muscular spasms and reduction of pain. Thus, the objective of this split mouth, randomized, blind, clinical trial will be to evaluate the postoperative period of 32 third molars in the patients from the São Paulo State University (Unesp), Institute of Science and Technology, São José dos Campos, Brasil. These evaluations will be performed on the third and seventh days after the extraction, where the patients will be analyzed by evaluator who will measure the edema, the opening of the mouth (evaluation of muscle spasm) and collect the pain table delivered in the immediate postoperative period, comparing thus, the benefit of therapeutic banding in the postoperative period of the extraction of lower third molars. The analogue pain scale (VAS), together with the Ustün et al. (2003) and the millimeter rule will be used to compare the data and the results will be submitted to descriptive statistics and compared by means of the statistical analysis of variance (ANOVA) and Tukey test with significance level of 5%.

DETAILED DESCRIPTION:
Extraction of third molars is the procedure of oral and maxillofacial surgery most commonly performed around the world, usually at the outpatient level. Its execution may result in the appearance of reversible and / or irreversible disorders, but the most observed signs and symptoms are pain, edema and trismus to a greater or lesser degree. Thus, there seems to be no consensus within the literature for a better type of post-surgical treatment that leads to less patient discomfort when undergoing this kind of surgery.

The objective of this randomized, blinded trial will be to evaluate the use of therapeutic bandaging, Therapy Tex ©, In reducing the signs and symptoms inherent to the postoperative period of the third molar extracts, semi-included or included .

The sample will consist of 32 lower third molars, semi-inclusively or included, divided into two groups simultaneously, namely:

Group I (16 teeth) - without therapeutic bandaging on face. Group II (16 teeth) - with therapeutic bandaging on face. The therapeutic bandaging method will be applied in the patients of group II, according to the previous randomization.The bandage will be applied immediately after surgery and before the end of the anesthetic effect. The skin should be cleaned with 70% alcohol in order to remove residue and oiliness, and then should be dried. If necessary, scrape the hairs of the region in which the tape will rest. The application of the bandage will be in the proposed regions using the "I" cutout, in which no additional trimming is made on the tape. The length may vary depending on the size of the patient's face. After being applied the bandage should be gently wiped to activate the acrylic components that generate adhesiveness and should remain on the face for 3 days.

The patient is asked to occlude, the dimension of the masseter muscle is determined by palpation. During palpation, point A is selected in the lower portion of the zygomatic arch and point B is close to the angle of the mandible. The tape will be placed along the direction of the muscle fibers.

Placement of the second tape will occur from the mandibular angle to the mental symphysis, accompanying the entire mandibular body in its medial portion covering the milo-hyoid muscles and the anterior belly of the digastric.

The results of the clinical evaluations will be submitted to descriptive statistics and compared by means of the statistical analysis of variance (ANOVA) and Tukey test with significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with need for extraction of third molars, regardless of gender;
2. Teeth in opposite hemiarches with similar positions;
3. Between 15 and 40 years of age;
4. That they agree to participate in the research voluntarily.

Exclusion Criteria:

1. Patients presenting with local or systemic alterations that contraindicate the procedure;
2. Use of anti-inflammatories in the last 15 days;
3. Third lower third molars in position and different inclusion classification on both sides;
4. Third erupted lower third molars.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-08-04 (Actual)

PRIMARY OUTCOMES:
Pain assessment | The scale will be provided on paper and divided into postoperative hours up to 3 days for the patient to note the degree of pain that varies between zero and ten
  Evaluated in patients in groups I and II. Scale of vas, with values from zero to ten, being zero without pain and ten the maximum of pain. This scale will be provided on paper and divided into postoperative hours up to 3 days.

SECONDARY OUTCOMES:
Edema assessment with a millimeter rule. | For investigators to measure facial edema, with pre and postoperative evaluations of 3 and 7 days
  Evaluated in patients in groups I and II. Used the method of Ustün et al. (2003) with a millimeter rule to obtain the measures.

OTHER OUTCOMES:
Trismus assessment with a millimeter rule. | To measure the buccal opening, the distance between the incisal edges of the maxillary and mandibular incisors, obtained with the patient sitting upright. Evaluated in the pre and postoperative periods of 3 and 7 days
  Evaluated in patients in groups I and II

CONTACTS AND LOCATIONS:
Overall Officials: Michelle B Moraes, PHD, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Michelle Bianchi de Moraes, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brignardello-Petersen R, Carrasco-Labra A, Araya I, Yanine N, Beyene J, Shah PS. Is adjuvant laser therapy effective for preventing pain, swelling, and trismus after surgical removal of impacted mandibular third molars? A systematic review and meta-analysis. J Oral Maxillofac Surg. 2012 Aug;70(8):1789-801. doi: 10.1016/j.joms.2012.01.008. Epub 2012 Mar 6. PMID 22398186
- [Result] UStun Y, Erdogan O, Esen E, Karsli ED. Comparison of the effects of 2 doses of methylprednisolone on pain, swelling, and trismus after third molar surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Nov;96(5):535-9. doi: 10.1016/S1079210403004645. PMID 14600686
- [Result] Maxwell C. Sensitivity and accuracy of the visual analogue scale: a psycho-physical classroom experiment. Br J Clin Pharmacol. 1978 Jul;6(1):15-24. doi: 10.1111/j.1365-2125.1978.tb01676.x. PMID 666944